CLINICAL TRIAL: NCT04872179
Title: International Prospective Registry of Patients With Alpha Thalassemia
Brief Title: International Registry of Patients With Alpha Thalassemia
Acronym: ATM Registry
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 16-21157-B
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Alpha-Thalassemia; Alpha Thalassemia Major; Alpha Thalassemia Minor
MeSH Terms: conditions — alpha-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an international prospective registry of patients with Alpha thalassemia to understand the natural history of the disease and the outcomes of fetal therapies, with the overall goal of improving the prenatal management of patients with Alpha thalassemia.

DETAILED DESCRIPTION:
The aim of this registry is to prospectively and retrospectively collect data on patients who are diagnosed with alpha thalassemia major and other alpha thalassemia mutations. Data collected will be used to:

1. Identify patient outcomes of therapies.
2. Improve clinical management of patients with ATM.
3. Improve medical decision making.
4. Improve quality of care.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of alpha thalassemia (prenatal or postnatal) with genotype consistent with ATM or BHFS phenotype
* referred to the University of California, San Francisco Fetal Treatment Center for fetal diagnosis, management and/or evaluation for the ongoing in utero stem cell transplantation clinical trial

Exclusion Criteria:

- none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be either self-enrolled, or enrolled through their prenatal provider (obstetrician, genetic counselor) or postnatal provider (hematologist, pediatrician).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2037-01 (Estimated)

PRIMARY OUTCOMES:
Survival to birth | 6 months
  Number of fetuses diagnosed with alpha thalassemia who survive to birth, compared to number of fetuses diagnosed with alpha thalassemia who have fetal demise or are terminated in utero. This is measured in number of fetuses alive at birth divided by number of all fetuses.
Vineland-3 Adaptive Behavior Scale | 10-15 years
  Results of neurodevelopmental testing using the Vineland Adaptive Behavior Scale version 3. The Vineland-3 scoring system is based on scores for three specific adaptive behavior domains: Communication, Daily Living Skills, and Socialization. The domain scores are expressed as standard scores with a mean of 100 and standard deviation of 15.

SECONDARY OUTCOMES:
Gestational age at birth | 6 months
  Gestational age of the child at birth. This is measured in weeks.
Mechanical ventilation | 1 year
  Duration (if any) of requiring mechanical ventilation after birth. This is measured in days.
Length of hospitalization | 6 months-1 year
  Duration of the child's hospitalization after birth. This is measured in days.
Resolution of hydrops | 6 months
  Evaluate whether receiving fetal therapy leads hydrops fetalis to resolve. This is measured by ultrasound findings.

CONTACTS AND LOCATIONS:
Overall Officials: Tippi C MacKenzie, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreger EM, Singer ST, Witt RG, Sweeters N, Lianoglou B, Lal A, Mackenzie TC, Vichinsky E. Favorable outcomes after in utero transfusion in fetuses with alpha thalassemia major: a case series and review of the literature. Prenat Diagn. 2016 Dec;36(13):1242-1249. doi: 10.1002/pd.4966. Epub 2016 Dec 7. PMID 27862048
- [Derived] Schwab ME, Lianoglou BR, Gano D, Gonzalez Velez J, Allen IE, Arvon R, Baschat A, Bianchi DW, Bitanga M, Bourguignon A, Brown RN, Chen B, Chien M, Davis-Nelson S, de Laat MWM, Ekwattanakit S, Gollin Y, Hirata G, Jelin A, Jolley J, Meyer P, Miller J, Norton ME, Ogasawara KK, Panchalee T, Schindewolf E, Shaw SW, Stumbaugh T, Thompson AA, Towner D, Tsai PS, Viprakasit V, Volanakis E, Zhang L, Vichinsky E, MacKenzie TC. The impact of in utero transfusions on perinatal outcomes in patients with alpha thalassemia major: the UCSF registry. Blood Adv. 2023 Jan 24;7(2):269-279. doi: 10.1182/bloodadvances.2022007823. PMID 36306387

DOCUMENTS (1):
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04872179/ICF_000.pdf